CLINICAL TRIAL: NCT06912451
Title: Sport Mouthguards: Devices for Preventing Dental and Alveolar Injuries in Sports - A Longitudinal Study
Brief Title: Sport Mouthguards: Devices for Preventing Dental Injuries in Sports
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio de Janeiro (FAPERJ) (Unknown)
Responsible Party: Principal Investigator, Mariana Pires da Costa, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 75456123.9.0000.0268
Record Dates: First submitted 2025-02-04; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Oral Health; Dental Trauma; Oral Health Knowledge, Attitude and Practice Among Patients; Mouth Protectors
Keywords: Mouth Protectors; Athletes; Sports; Dental Trauma; Questionnaire; Oral health
MeSH Terms: conditions — Behavior | interventions — Mouth Protectors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sport Mouthguard (Experimental): After the initial consultation for clinical examination data collection and anamnesis, an impression of the patient's upper dental arch will be made to create a custom mouthguard. This mouthguard will be made using two 3mm vinyl acetate ethylene sheets, following the recommendations for an appropriate mouthguard regarding trauma prevention and patient comfort.
  Interventions: Device: Sport custom mouthguard

INTERVENTIONS:
Device: Sport custom mouthguard — This mouthguard will be made using two 3mm vinyl acetate ethylene sheets in a vacuum machine, following the recommendations for an appropriate mouthguard regarding trauma prevention and patient comfort. The patients will be monitored after 1, 3, and 6 months of using the mouthguard.
  Other Names: Mouthguard; Mouth Protector

SUMMARY:
Objective: To evaluate the impact of mouthguards (MG) on acceptability, incidence of soft tissue injuries, periodontal and salivary parameters, as well as on the perception of the body in sports practice (PeCoPes) and on the quality of life of athletes, and evaluate the consequences of use on the characteristics, state of conservation, and biological and physical properties of the MG itself. Methodology: This is a longitudinal study that will include children, adolescents, and adults aged 7 to 30 years who practice sports and require MGs. Sociodemographic data, medical history, dental history, dietary habits, and sports practice data will be collected. Participants will undergo a complete oral clinical examination. Data on knowledge of traumatic dental injuries (TDI) and MGs will also be collected. Before the MG is delivered, immediately after installation, and at 1, 3, and 6 months after use, the following parameters will be evaluated: presence of mucosal injuries, visible plaque index, gingival bleeding index, salivary flow, salivary pH, buffering capacity, and salivary microorganism count. Acceptability will be evaluated before the MG is delivered, immediately after delivery, and at 1, 3, and 6 months after use. PeCoPes and quality of life will be assessed before, 1, 3, and 6 months after MG use. The MG will be evaluated for bacterial contamination, delamination, roughness, dimensional changes related to shape and thickness, color change, and conservation status. The data will be tabulated and analyzed using SPSS 21.0, and appropriate statistical tests (p<0.05) will be performed according to the study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents, and adults aged 7 to 30 years, with no systemic health issues, of both genders;
* Engaging in sports practice at least twice a week.

Exclusion Criteria:

* Presence of cavitated dental caries and/or periodontitis;
* Angle Class III malocclusion with negative anterior overjet;
* Presence of non-removable prostheses or any other accessory in the upper or lower arch that may interfere with the adaptation of the mouthguard;
* Use of medications that may interfere with any salivary parameters;
* Children, adolescents, and adults with neurological disorders or communication difficulties.

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Acceptability will be evaluated before the MG is delivered, immediately after delivery, and at 1, 3, and 6 months after use.
  Acceptability will be assessed through a questionnaire on changes in the oral cavity associated with the use of the MG or in the MG itself. This questionnaire was developed by the authors of the study.
Incidence of soft tissue injuries | Before the MG is delivered, and at 1, 3, and 6 months after use
  The following parameter will be evaluated: presence of mucosal injuries through clinical examinations
Periodontal and salivary parameters | Before the MG is delivered, immediately after installation, and at 1, 3, and 6 months after use.
  The following parameters will be evaluated: visible plaque index, gingival bleeding index, salivary flow, salivary pH, buffering capacity, and salivary microorganism count.

SECONDARY OUTCOMES:
The perception of the body in sports practice (PeCoPes) | PeCoPes will be assessed before, 1, 3, and 6 months after MG use.
  The perception of the body in sports practice (PeCoPes) will be assessed through a previously validated questionnaire.
The quality of life of athletes | Quality of life will be assessed before, 1, 3, and 6 months after MG use.
  The quality of life will be assessed through some previously validated questionnaires.
The consequences of use on the characteristics, state of conservation, and biological and physical properties of the MG itself. | Before the MG is delivered, immediately after installation, and at 1, 3, and 6 months after use.
  The MG will be evaluated for bacterial contamination, delamination, roughness, dimensional changes related to shape and thickness, color change, and conservation status.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The results will be released after the completion of the longitudinal study, which forms part of the responsible reseacher's PhD thesis.